CLINICAL TRIAL: NCT01188512
Title: A Phase 1, Single Centre, Dose-escalating, Placebo-controlled Study of a Genetically Modified B. Pertussis Strain Given as a Single Intranasal Dose to Healthy Adult Male Volunteers
Brief Title: First Adult Safety Trial on Nasal Live Attenuated B. Pertussis Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: European Union (Other); Swedish Institute for Infectious Disease Control (Other); Innogenetics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BT06-04; 2010-019936-11 (EudraCT Number)
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2012-01

CONDITIONS: Pertussis
Keywords: Live nasal vaccine for prevention of pertussis
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BPZE1 - Low dose (Experimental): 1,000 colony forming units (cfu) of BPZE1
  Interventions: Biological: BPZE1
- BPZE1- middle dose (Experimental): 100,000 colony forming units (cfu) of BPZE1
  Interventions: Biological: BPZE1
- BPZE1 - High dose (Experimental): 10,000,000 colony forming units (cfu) of BPZE1
  Interventions: Biological: BPZE1
- Placebo (Placebo Comparator): Formulation buffer
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BPZE1 — Individuals will be vaccinated once intranasally with the designated dose of BPZE1 Dose 2 x 0.1 mL (0.1 mL per nostril).
  Arms: BPZE1 - High dose; BPZE1 - Low dose; BPZE1- middle dose
Biological: Placebo — Individuals will get placebo once intranasally. Dose 2 x 0.1 mL (0.1 mL per nostril).
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a new live attenuated vaccine against whooping-cough. It is a phase1, single centre, dose-escalating, placebo-controlled study on a genetically modified B. pertussis strain given as a single intranasal dose to healthy adult male volunteers.

Effective vaccines are needed to protect young infants (from 0 to 6 months, today the most vulnerable age group), preferably after a single administration very early in life. The successful outcome of this project would constitute an important milestone towards nasal vaccination of infants, possibly at birth with a novel, single-dose pertussis vaccine. Our ultimate aim is to protect infants in the most vulnerable age group, before the regular vaccination schedule using already available vaccines is applied. The ultimate aim is thus not to replace current vaccination schedules with available vaccines, but to add a first nasal vaccination to protect very early in life.

ELIGIBILITY:
Inclusion Criteria:

Subject will be included in the study if he meets all the following criteria:

* Healthy male born between 1979 and 1991 who has not experienced clinical pertussis (lab. Verified) during the past 10 years and who has not been vaccinated with any pertussis vaccine.
* Informed consent form signed by the subject.
* Subject shall be able to attend all scheduled visits and to understand and comply with the study procedures (e.g. able to read and write Swedish).

Exclusion Criteria:

If any of the following criteria are met, the subject must not be included in the study:

* Individuals with pertussis toxin serum IgG antibodies ≥20 units/mL.
* Blood pressure after resting ≥ 150/90 mmHg.
* Heart rate after resting ≥80 bpm.
* Respiratory rate after resting ≥ 20/minute.
* Unwillingness to refrain from the use of nicotine products from screening through day 28.
* Use of narcotic drugs/alcohol and/or a history of previous use of drug/alcohol abuse whitin the past 2 years prior to screening
* The subject has donated blood or suffered from blood loss of at least 450 ml (1 unit of blood) within 60 days prior to screening or donated plasma within 14 days prior to screening.
* Receipt of immunoglobulin, blood derived products, systemic corticosteroids or other immunosuppressant drugs within 90 days prior to day 0.
* Use of corticosteroids in the respiratory tract(e.g. nasal steroids, inhaled steroids) whitin 30 days prior to day 0.
* Use of herbal medications or dietary supplements within 7 days prior to day 0 at the discretion of the investigator. Unwillingness to refrain from herbal medications or dietary supplements within 30 days after day 0 at the discretion of the investigator.
* Receipt of a vaccine within the last 30 days prior to day 0 or planned vaccination within the next 30 days after day 0.
* Evolving encephalopathy not attributable to another identifiable cause within 7 days of administration of a previous dose of any vaccine.
* Known hypersensitivity to any component of the study vaccine.
* Current participation in any other clinical trial or participation (and during the whole study) in any clinical trial in the previous 3 months prior to day 0.
* Inability to adhere to the protocol, including plans to move from the area.
* Family history of congenital or hereditary immunodeficiency (first degree).
* Infection with HIV, hepatitis B or C.
* Any medical condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* Clinically significant abnormal laboratory values at the discretion of the investigator.
* Person in frequent contact with children less than 1 year of age (father, childcare worker, nurse, etc…) or residence in the same household as persons with known immunodeficiency.

Ages: 19 Years to 31 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
General safety and local tolerability in the respiratory tract of a single ascending dose of the genetically modified B. pertussis strain | 6 months
  To determine
  * general safety, i. e. general well-being of the volunteers and any symptoms felt by the volunteers with onset within one month after vaccine administration.
  * vital signs: Blood pressure, heart rate, respiratory rate, oral temperature.
  * abnormalities in the following laboratory data: Haemoglobin, total and differential white blood cell count, platelets (thrombocytes).
  * specific side effects: Local symptoms from the respiratory tract: Sneezing, swollen nose, cough, bleeding from the nose, pain or other symptoms from the ear, symptoms from the eyes (redness, secretion).

SECONDARY OUTCOMES:
Attachment of the BPZE1 strain to the nasopharyngeal mucosa | Up to 50 days after vaccination
  Detection of colonizing BPZE1 bacteria in nasopharyngeal culture
Immunogenicity | 6 months
  Immune responses will be determined by serum IgG and IgA, IgG and IgA in saliva and nasopharyngeal aspirate, cytokines and numbers of effector and memory T and B cells after stimulation with the various B. pertussis antigens.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Locht, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Nabil Al-Tawil, MD, PhD, Principal Investigator — Karolinska Trial Alliance; Rigmor Thorstensson, PhD, Principal Investigator — Swedish Institute for Infectious Disease Control
Locations (1):
- Karolinska University Hospital, Solna, Sweden

REFERENCES:
- [Background] Mielcarek N, Debrie AS, Raze D, Bertout J, Rouanet C, Younes AB, Creusy C, Engle J, Goldman WE, Locht C. Live attenuated B. pertussis as a single-dose nasal vaccine against whooping cough. PLoS Pathog. 2006 Jul;2(7):e65. doi: 10.1371/journal.ppat.0020065. PMID 16839199
- [Background] Feunou PF, Ismaili J, Debrie AS, Huot L, Hot D, Raze D, Lemoine Y, Locht C. Genetic stability of the live attenuated Bordetella pertussis vaccine candidate BPZE1. Vaccine. 2008 Oct 23;26(45):5722-7. doi: 10.1016/j.vaccine.2008.08.018. Epub 2008 Aug 30. PMID 18762220
- [Background] Mielcarek N, Debrie AS, Mahieux S, Locht C. Dose response of attenuated Bordetella pertussis BPZE1-induced protection in mice. Clin Vaccine Immunol. 2010 Mar;17(3):317-24. doi: 10.1128/CVI.00322-09. Epub 2010 Jan 27. PMID 20107007
- [Background] Kavanagh H, Noone C, Cahill E, English K, Locht C, Mahon BP. Attenuated Bordetella pertussis vaccine strain BPZE1 modulates allergen-induced immunity and prevents allergic pulmonary pathology in a murine model. Clin Exp Allergy. 2010 Jun;40(6):933-41. doi: 10.1111/j.1365-2222.2010.03459.x. Epub 2010 Feb 22. PMID 20184606
- [Background] Skerry CM, Cassidy JP, English K, Feunou-Feunou P, Locht C, Mahon BP. A live attenuated Bordetella pertussis candidate vaccine does not cause disseminating infection in gamma interferon receptor knockout mice. Clin Vaccine Immunol. 2009 Sep;16(9):1344-51. doi: 10.1128/CVI.00082-09. Epub 2009 Jul 22. PMID 19625486
- [Result] Thorstensson R, Trollfors B, Al-Tawil N, Jahnmatz M, Bergstrom J, Ljungman M, Torner A, Wehlin L, Van Broekhoven A, Bosman F, Debrie AS, Mielcarek N, Locht C. A phase I clinical study of a live attenuated Bordetella pertussis vaccine--BPZE1; a single centre, double-blind, placebo-controlled, dose-escalating study of BPZE1 given intranasally to healthy adult male volunteers. PLoS One. 2014 Jan 8;9(1):e83449. doi: 10.1371/journal.pone.0083449. eCollection 2014. PMID 24421886
- [Result] Jahnmatz M, Amu S, Ljungman M, Wehlin L, Chiodi F, Mielcarek N, Locht C, Thorstensson R. B-cell responses after intranasal vaccination with the novel attenuated Bordetella pertussis vaccine strain BPZE1 in a randomized phase I clinical trial. Vaccine. 2014 Jun 5;32(27):3350-6. doi: 10.1016/j.vaccine.2014.04.048. Epub 2014 Apr 29. PMID 24793938
- [Derived] Schnoeller C, Roux X, Sawant D, Raze D, Olszewska W, Locht C, Openshaw PJ. Attenuated Bordetella pertussis vaccine protects against respiratory syncytial virus disease via an IL-17-dependent mechanism. Am J Respir Crit Care Med. 2014 Jan 15;189(2):194-202. doi: 10.1164/rccm.201307-1227OC. PMID 24261996